CLINICAL TRIAL: NCT04331977
Title: Effectiveness of Two Rapid Maxillary Expanders (Quadhelix vs Hyrax) in Improving the Transverse Skeletal and Dental Dimensions in Patients With Cleft Lip and Palate: A Randomized Clinical Trial
Brief Title: Effectiveness of Two Maxillary Expanders in Improving the Transverse Skeletal and Dental Dimensions in Patients With Cleft Lip and Palate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abd El-Ghafour, Lecturer of Orthodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 121
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Cleft Lip and Palate; Maxillary Expansion
MeSH Terms: conditions — Cleft Lip | interventions — Palatal Expansion Technique

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadhelix Group (Experimental)
  Interventions: Device: Maxillary Expansion
- Hyrax Group (Active Comparator)
  Interventions: Device: Maxillary Expansion

INTERVENTIONS:
Device: Maxillary Expansion — 2 appliances to expand the maxillary arch

SUMMARY:
This randomized controlled trial is designed to compare between quadlelix appliance vs hyrax expander regrading the their effectiveness in maxillary expansion in patients with cleft.

ELIGIBILITY:
Inclusion Criteria:

* Mixed dentition stage;
* Both males and females;
* Lip repair performed between 3 and 6 months of age and palate repair performed between 12 and 24 months of age;
* Presence of maxillary constriction and posterior crossbite and need for maxillary expansion previous to the secondary bone graft;
* Permanent first maxillary molars present;
* Good periodontal health;
* No previous orthodontic treatment; and

Exclusion Criteria:

* Presence of a syndrome in companion with the present cleft defect.
* Previous secondary alveolar bone grafting.
* Taking medications affecting growth.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Maxillary Expansion | 6 months
  Amount of Maxillary Expansion to be measured as distances (mm) on CBCTs and dental models.
Maxillary Expansion | 6 months
  mount of Maxillary Expansion to be measured as angles (degrees) on CBCTs and dental models.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided